CLINICAL TRIAL: NCT04517331
Title: Comparison of Single and Double Injection Ultrasound-Guided Bilateral Thoracic Paravertebral Block Effects in Patients Undergoing Reduction Mammaplasty: A Prospective Randomized Controlled Study
Brief Title: Single and Double Injection Bilateral Thoracic Paravertebral Blocks in Reduction Mammaplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emine Aysu Salviz, MD, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2016/1282
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Pain, Postoperative
Keywords: Thoracic paravertebral blocks; Postoperative analgesia, numeric rating scale; Dermatomal blockade distribution; Postoperative time until first pain; Analgesic consumption; Reduction mammaplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients undergoing reduction mammaplasty, received single or double injection bilateral thoracic paravertebral block (TPVB) for postoperative analgesia
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: * All TPVB procedures were performed by the same 3 senior anesthesiology residents, always under the supervision of 2 attending anesthesiologists (1 senior resident with 1 attending anesthesiologist at a time)
  * Preoperatively, the anesthesiologists who were blinded to the group of that specific patient evaluated the sensorial blockade of dermatomes separately on both sides
  * Postoperatively, different anesthesiologists who did not participate in the TPVB performance process of that specific patient and were totally blinded to the group again collected the data.
  * Surgeons were also blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (single injection TPVB group) (Active Comparator): Patients received bilateral single injection ultrasound-guided TPVB at the level of T3-T4 with 20 mL bupivacaine 0.375% per injection/side.
  Interventions: Procedure: Thoracic paravertebral block-single injection
- Group D (double injection TPVB group) (Active Comparator): Patients received bilateral double injection ultrasound-guided TPVB at the level of T2-T3 and T4-T5 with 10 mL bupivacaine 0.375% per injection (20 mL bupivacaine 0.375% per side as the single injection group).
  Interventions: Procedure: Thoracic paravertebral block-double injection

INTERVENTIONS:
Procedure: Thoracic paravertebral block-single injection — The blocks were performed at the T3-T4 level bilaterally to block the dermatomes between the T2 and T6 levels (breast innervation area).
  Arms: Group S (single injection TPVB group)
Procedure: Thoracic paravertebral block-double injection — The blocks were performed at both T2-T3 and T4-T5 levels bilaterally to block the dermatomes between the T2 and T6 levels (breast innervation area).
  Arms: Group D (double injection TPVB group)

SUMMARY:
This study compares the analgesic effects and dermatomal blockade distributions of single and double injection bilateral thoracic paravertebral block (TPVB) techniques in patients undergoing reduction mammaplasty.

After obtaining ethics committee approval; 60 patients scheduled for elective bilateral reduction mammoplasty and gave written informed consent, were included in the study. The patients were randomized in one of single (Group S: T3-T4) or double injections (Group D: T2-T3&T4-T5) bilateral TPVB groups (bupivacaine 0.375% 20 mL per side). All patients' dermatomal blockade distributions (T2-T6) were followed for 30 minutes, and then they were given general anesthesia. Before extubation, 1 g IV paracetamol was applied to all. Postoperatively, patients in both groups received IV paracetamol 1 g when numeric rating scale (NRS) pain score ≥4, and also tramadol 1 mg/kg if they defined NRS≥4 again after 1 h. The primary endpoint was NRS pain scores at postoperative 12th hour. The secondary endpoints were NRS scores and dermatomal blockade distributions through the postoperative first 48 hours, postoperative time until first pain, the total numbers of analgesic requirements on days 1 and 2.

DETAILED DESCRIPTION:
This prospective randomized controlled study compares the analgesic effects and dermatomal blockade distributions of single and double injection bilateral thoracic paravertebral block (TPVB) techniques in patients undergoing reduction mammaplasty.

After obtaining ethics committee approval; 60 patients scheduled for elective bilateral reduction mammoplasty and gave written informed consent, were included in the study. The inclusion criteria were female gender, aging between 18 and 70 years, American Society of Anesthesiologists (ASA) physical status of 1-3, capable of consenting, understanding the instructions for using the NRS pain scores and replying the study-based questions, lack of contraindications to regional anesthesia (allergy to a LA, local infection, and coagulopathy) and especially TPVB, absence of mental/psychiatric disorders, chronic analgesic/opioid use and alcohol/illicit drug use. The patients were randomized in one of single (Group S: T3-T4-bupivacaine 0.375% 20 mL/injection) or double injections (Group D: T2-T3&T4-T5-bupivacaine 0.375% 10 mL/injection) bilateral TPVB groups using the sealed envelopes technique. All patients' dermatomal (sensorial) blockade distributions (T2-T6) were tested bilaterally between T2 and T6 dermatomal levels on the midclavicular line in every 5 minutes through the first 30 minutes after TPVB performances, by using the pin-prick test, and then they were given standard general anesthesia. Before extubation, 1 g IV paracetamol was applied to all. The NRS pain scores (0: no pain and 10: worst pain imaginable), and the dermatomal blockade distribution/numbers of blocked dermatomes of all patients on both sides were asked and documented on postoperative 0th min, 1st, 2nd, 6th, 12th, 24th and 48th hours. Postoperatively, patients in both groups received IV paracetamol 1 g when NRS pain score ≥4, and also tramadol 1 mg/kg if they defined NRS≥4 again after 1 h. The primary endpoint was NRS pain score at 12th hour. The secondary endpoints included the NRS pain scores and the dermatomal blockade distribution/numbers of blocked dermatomes through the postoperative first 48 hours, block application times, number of patients experienced hypotension or required fentanyl intraoperatively, length of stay in postoperative care unit (PACU), postoperative time until first pain (NRS≥4), the total numbers of paracetamol and tramadol requirements, incidence of postoperative nausea and vomiting (PONV) and duration of sleep on postoperative days 1 and 2, patient and surgeon satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status of 1-3
* Capable of consenting
* Capable of understanding the instructions for using the NRS pain scores
* Capable of replying the study-based questions
* Lack of contraindications to regional anesthesia (allergy to a LA, local infection, and coagulopathy) and especially TPVB
* Absence of mental/psychiatric disorders
* Absence of chronic analgesic/opioid use
* Absence of alcohol/illicit drug use

Exclusion Criteria:

* Patient refusal
* American Society of Anesthesiologists (ASA) physical status of 4
* Not capable of consenting
* Not capable of understanding the instructions for using the NRS pain scores
* Not capable of replying the study-based questions
* Contraindications to regional anesthesia (allergy to a LA, local infection, and coagulopathy) and especially TPVB
* Presence of mental/psychiatric disorders
* Presence of chronic analgesic/opioid use
* Presence of alcohol/illicit drug use

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Pain (Numeric rating scale (NRS)) score | 12th hour
  NRS pain score (0: no pain, 10: worst pain imaginable) on postoperative 12th hour

SECONDARY OUTCOMES:
Pain (Numeric rating scale (NRS)) score | 0-48 hours
  NRS pain scores (0: no pain, 10: worst pain imaginable) on postoperative 0th min, 1st, 2nd, 6th, 24th and 48th hours on both sides
Dermatomal blockade distribution/numbers of blocked dermatomes | 0-30 minutes
  Preoperatively, the sensorial blockade was tested bilaterally between the T2 and T6 dermatomal levels (4 regions) on the midclavicular line of the patients in every 5 min through the first 30 min after TPVB performances, by using the pin-prick test. Sensations: "normal", "decreased sensation" or "total anesthesia" separately on both sides. The answers such as "decreased sensation" or "total anesthesia" in different dermatomal regions within T2-T6 were accepted as "successfully blocked dermatome", and the numbers of blocked dermatomes out of 4 dermatomal regions were noted for the right and the left sides.
Dermatomal blockade distribution/numbers of blocked dermatomes | 0-48 hours
  Postoperatively, the sensorial blockade was tested bilaterally between the T2 and T6 dermatomal levels (4 regions) on the midclavicular line of the patients on postoperative 0th min, 1st, 2nd, 6th, 12th, 24th and 48th hours, by using the pin-prick test. Sensations: "normal", "decreased sensation" or "total anesthesia" separately on both sides. The answers such as "decreased sensation" or "total anesthesia" in different dermatomal regions within T2-T6 were accepted as "successfully blocked dermatome", and the numbers of blocked dermatomes out of 4 dermatomal regions were noted for the right and the left sides.
Block application time | 2-20 minutes
  The bilateral TPVB application time was defined as the time period between the needle insertion at the first determined level and the needle withdrawal from the last determined level.
Number of patients experienced hypotension intraoperatively | Intraoperative 2-4 hours
  The mean arterial pressure (MAP) decreased >20% below preinduction value
Number of patients required fentanyl intraoperatively | Intraoperative 2-4 hours
  If a ≥ 20% increase above preinduction values in MAP or HR was observed during the perioperative period, additional fentanyl dose (1 µg/kg) was applied intravenously.
Length of stay in postoanesthesia care unit (PACU) | 0-1 hours
  Discharge from PACU was determined using the White Fast tracking score ≥12, whereas none of the parameters was <1 in any category
Postoperative time until first pain | 0-48 hours
  Postoperative first pain description (NRS ≥4)
Paracetamol consumption/the total numbers of paracetamol requirements | 0-48 hours
  Paracetamol was used when postoperative pain NRS ≥4 in the postanesthesia care unit or on the wards (on postoperative days 1 and 2)
Tramadol consumption/the total numbers of tramadol requirements | 0-48 hours
  Tramadol was used when postoperative pain NRS ≥4 again after 1 h of paracetamol application in the postanesthesia care unit or on the wards (on postoperative days 1 and 2)
Incidence of postoperative nausea and vomiting (PONV) | 0-48 hours
  Number of feeling nausea or vomiting (on postoperative days 1 and 2)
Duration of sleep | 0-48 hours
  Total hours of sleep per day (on postoperative days 1 and 2)
Patient satisfaction | 0-48 hours
  Satisfaction score: 0: very unsatisfied, 3: very satisfied
Surgeon satisfaction | 0-48 hours
  Satisfaction score: 0: very unsatisfied, 3: very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Emine A Salviz, MD,AssocProf, Principal Investigator — Study Principal Investigator, Corresponding author
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salviz EA, Sivrikoz N, Ozonur A, Orhan-Sungur M, Savran-Karadeniz M, Altun D, Hocaoglu E, Celet-Ozden B, Tugrul KM. Ultrasound-Guided Bilateral Thoracic Paravertebral Blocks as an Adjunct to General Anesthesia in Patients Undergoing Reduction Mammaplasty: A Historical Cohort Study. Plast Reconstr Surg. 2017 Jan;139(1):20e-28e. doi: 10.1097/PRS.0000000000002842. PMID 28027224
- [Result] Kaya FN, Turker G, Mogol EB, Bayraktar S. Thoracic paravertebral block for video-assisted thoracoscopic surgery: single injection versus multiple injections. J Cardiothorac Vasc Anesth. 2012 Feb;26(1):90-4. doi: 10.1053/j.jvca.2011.09.008. Epub 2011 Nov 4. PMID 22055006
- [Result] Kaya FN, Turker G, Basagan-Mogol E, Goren S, Bayram S, Gebitekin C. Preoperative multiple-injection thoracic paravertebral blocks reduce postoperative pain and analgesic requirements after video-assisted thoracic surgery. J Cardiothorac Vasc Anesth. 2006 Oct;20(5):639-43. doi: 10.1053/j.jvca.2006.03.022. Epub 2006 Aug 8. PMID 17023279